CLINICAL TRIAL: NCT02049736
Title: The Effect of Telbivudine on Renal Function and Proteinuria in Patients With Chronic Hepatitis B Infection and Chronic Kidney Diseases
Brief Title: Effect of Telbivudine on Renal Function and Proteinuria in Patients With CHB & Chronic Renal Diseases
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit patients
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Henry LY Chan, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Telbivudine for CKD
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telbivudine (Experimental)
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Drug: Telbivudine

SUMMARY:
Chronic kidney disease (CKD) and chronic viral hepatitis due to hepatitis B virus (HBV) are both major public health problems. Treatment of chronic HBV infection in CKD patients, however, is not well defined because of insufficient data from clinical trials. Telbivudine is a new antiviral that provides effective and sustained viral suppression in patients with compensated chronic hepatitis B infection. Unlike other nucleotide and nucleoside analogues, renal toxicity is uncommon in telbivudine, and dosage adjustment is not required in patients with mild renal impairment. We propose to conduct an open-label single-arm study to evaluate the effect of telbivudine on renal function and proteinuria in patients with chronic HBV infection and mild-to-moderate renal impairment. Twenty patients with chronic HBV infection and chronic kidney disease (estimated glomerular filtration rate 15 to 60 ml/min) will be recruited. They will be treated with telbivudine, with the dosage adjusted according to thei renal function, for 5 years. Serum HBV DNA, proteinuria, renal function, and urinary inflammatory markers will be monitored.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major public health problem worldwide over the past few decades, partly because of the increasing prevalence of hypertension, diabetes mellitus, and elderly individuals in most countries. In southeast Asia, chronic viral hepatitis due to hepatitis B virus (HBV) also poses significant morbidity and mortality [2]. Chronic HBV infection can cause chronic glomerulonephritis and CKD. More importantly, patients with CKD, irrespective to the underlying renal diagnosis, who acquire HBV infection have higher morbidity and mortality rates, and the management of chronic HBV infections among CKD patients with antiviral agents is associated with a high risk of adverse effects. The optimal management of CKD associated with chronic HBV infection is not well defined because of insufficient data from clinical trials.

Telbivudine (Sebivo®; Tyzeka®) is a synthetic nucleoside analogue that inhibits replication of HBV. Telbivudine is a potent antiviral that provides effective and sustained viral suppression in patients with compensated chronic hepatitis B infection, and is used in the treatment of adults with chronic hepatitis B with evidence of viral replication and persistently elevated serum transaminase levels, or histological evidence of active disease. Unlike most of the other nucleoside and nucleotide analogues, renal toxicity of telbivudine is uncommon, and dose adjustment is only necessary for patients with moderate to severe renal impairment. Recent data further suggest that telbivudine treatment may have a beneficial effect on renal function.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years
* hepatitis B surface antigen (HBsAg) positive
* clinical indication for antiviral therapy according to the Asian Pacific guideline [16]
* HBeAg positive, ALT >2 times upper limit of normal AND HBV DNA >20,000 IU/ml AND HBV DNA <9 log10 copies/mL; OR
* HBeAg negative, ALT >2 times upper limit of normal AND HBV DNA >2,000 IU/ml AND HBV DNA <7 log10 copies/mL; OR
* Evidence of advanced liver fibrosis or liver cirrhosis AND detectable HBV DNA
* estimated glomerular filtration rate (GFR) 15 to 60 ml/min/1.73m2
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* Pregnancy, lactating or childbearing potential without effective method of birth control
* Severe gastrointestinal disorders that interfere with their ability to receive or absorb oral medication
* History of malignancy, including leukemia and lymphoma within the past 2 years
* Active systemic infection.
* Any other severe coexisting disease such as, but not limited to, advanced liver cirrhosis, myocardial infarction, cerebrovascular accident, malignant hypertension
* History of drug or alcohol abuse within past 2 years
* Patients receiving antiviral therapy for chronic hepatitis B within the past 12 months
* Patients receiving treatment of corticosteroid or other immunosuppressive / cytotoxic agents
* On other investigational drugs within last 3 months
* History of a psychological illness or condition such as to interfere with the patient's ability to understand the requirement of the study
* History of non-compliance
* Known history of sensitivity or allergy to telbivudine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change in estimated glomerular filtration rate | every 3 months for 5 years

SECONDARY OUTCOMES:
proteinuria | every 3 months for 5 years
HBV DNA level | every 6 months for 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Suen Man Shook Hepatitis Center, Institute of Digestive Disease, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Coresh J, Byrd-Holt D, Astor BC, Briggs JP, Eggers PW, Lacher DA, Hostetter TH. Chronic kidney disease awareness, prevalence, and trends among U.S. adults, 1999 to 2000. J Am Soc Nephrol. 2005 Jan;16(1):180-8. doi: 10.1681/ASN.2004070539. Epub 2004 Nov 24. PMID 15563563
- [Background] Chen J, Wildman RP, Gu D, Kusek JW, Spruill M, Reynolds K, Liu D, Hamm LL, Whelton PK, He J. Prevalence of decreased kidney function in Chinese adults aged 35 to 74 years. Kidney Int. 2005 Dec;68(6):2837-45. doi: 10.1111/j.1523-1755.2005.00757.x. PMID 16316361
- [Background] Bhimma R, Coovadia HM. Hepatitis B virus-associated nephropathy. Am J Nephrol. 2004 Mar-Apr;24(2):198-211. doi: 10.1159/000077065. Epub 2004 Feb 25. PMID 14988643
- [Background] Chacko EC, Surrun SK, Mubarack Sani TP, Pappachan JM. Chronic viral hepatitis and chronic kidney disease. Postgrad Med J. 2010 Aug;86(1018):486-92. doi: 10.1136/pgmj.2009.092775. PMID 20709771
- [Background] Wong PN, Fung TT, Mak SK, Lo KY, Tong GM, Wong Y, Loo CK, Lam EK, Wong AK. Hepatitis B virus infection in dialysis patients. J Gastroenterol Hepatol. 2005 Nov;20(11):1641-51. doi: 10.1111/j.1440-1746.2005.03837.x. PMID 16246180
- [Background] London WT, Drew JS, Lustbader ED, Werner BG, Blumberg BS. Host responses to hepatitis B infection in patients in a chronic hemodialysis unit. Kidney Int. 1977 Jul;12(1):51-8. doi: 10.1038/ki.1977.78. PMID 894916
- [Background] Peters MG. Special populations with hepatitis B virus infection. Hepatology. 2009 May;49(5 Suppl):S146-55. doi: 10.1002/hep.22965. PMID 19399810
- [Background] Girndt M, Kohler H. Hepatitis B virus infection in hemodialysis patients. Semin Nephrol. 2002 Jul;22(4):340-50. PMID 12118399
- [Background] Fabrizi F, Messa P, Basile C, Martin P. Hepatic disorders in chronic kidney disease. Nat Rev Nephrol. 2010 Jul;6(7):395-403. doi: 10.1038/nrneph.2010.37. Epub 2010 Apr 13. PMID 20386560
- [Background] McKeage K, Keam SJ. Telbivudine: a review of its use in compensated chronic hepatitis B. Drugs. 2010 Oct 1;70(14):1857-83. doi: 10.2165/11204330-000000000-00000. PMID 20836578
- [Background] But DY, Yuen MF, Fung J, Lai CL. Safety evaluation of telbivudine. Expert Opin Drug Saf. 2010 Sep;9(5):821-9. doi: 10.1517/14740338.2010.507190. PMID 20662545
- [Background] Zhou XJ, Swan S, Smith WB, Marbury TC, Dubuc-Patrick G, Chao GC, Brown NA. Pharmacokinetics of telbivudine in subjects with various degrees of renal impairment. Antimicrob Agents Chemother. 2007 Dec;51(12):4231-5. doi: 10.1128/AAC.00557-07. Epub 2007 Sep 17. PMID 17875994
- [Background] Lai CL, Gane E, Liaw YF, Hsu CW, Thongsawat S, Wang Y, Chen Y, Heathcote EJ, Rasenack J, Bzowej N, Naoumov NV, Di Bisceglie AM, Zeuzem S, Moon YM, Goodman Z, Chao G, Constance BF, Brown NA; Globe Study Group. Telbivudine versus lamivudine in patients with chronic hepatitis B. N Engl J Med. 2007 Dec 20;357(25):2576-88. doi: 10.1056/NEJMoa066422. PMID 18094378
- [Background] Gane EJ, Wang Y, Liaw YF, Hou J, Thongsawat S, Wan M, Moon YM, Jia J, Chao YC, Niu J, Leung N, Samuel D, Hsu CW, Bao W, Lopez P, Avila C. Efficacy and safety of prolonged 3-year telbivudine treatment in patients with chronic hepatitis B. Liver Int. 2011 May;31(5):676-84. doi: 10.1111/j.1478-3231.2011.02490.x. Epub 2011 Mar 16. PMID 21457439
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Szeto CC, Chow KM, Kwan BC, Chung KY, Leung CB, Li PK. Oral calcitriol for the treatment of persistent proteinuria in immunoglobulin A nephropathy: an uncontrolled trial. Am J Kidney Dis. 2008 May;51(5):724-31. doi: 10.1053/j.ajkd.2007.12.038. Epub 2008 Apr 3. PMID 18436082
- [Background] Grubb A, Nyman U, Bjork J, Lindstrom V, Rippe B, Sterner G, Christensson A. Simple cystatin C-based prediction equations for glomerular filtration rate compared with the modification of diet in renal disease prediction equation for adults and the Schwartz and the Counahan-Barratt prediction equations for children. Clin Chem. 2005 Aug;51(8):1420-31. doi: 10.1373/clinchem.2005.051557. Epub 2005 Jun 16. PMID 15961546